CLINICAL TRIAL: NCT02787915
Title: DC1s-CTL Cell Therapy to Treat Patients With Renal Cell Carcinoma After Radical Resection
Brief Title: DC1s-CTL Cellular Therapy for Renal Cell Carcinoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, Junnian Zheng, professor, Xuzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XYFY2016-KL012-01
Record Dates: First submitted 2016-05-26; First posted 2016-06-01 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2016-05

CONDITIONS: Renal Cell Carcinoma
Keywords: dendritic cells; cytotoxic T lymphocyte; DC vaccine
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- dendritic cell vaccine (Experimental): DC1-CTL cellular therapy
  Interventions: Biological: DC1-CTL

INTERVENTIONS:
Biological: DC1-CTL — Autologous cytotoxic of T lymphocytes (CTL) were induced by type-1 polarized dendritic cells (DC1) loaded with MAGE-3/MAGE-4/survivin/ her2 /COX-2 CTL epitope peptides .

SUMMARY:
This trial is to evaluate the safety and effectiveness of autologous type-1 polarized dendritic cell vaccines (patients' autologous DC1s loaded with multiple antigens CTL epitope peptide complexes), after radical resection for patients with stage III-IV renal cell carcinoma. Autologous cytotoxic of T lymphocytes (CTL) induced by type-1 polarized dendritic cells (DC1) loaded with MAGE-3/MAGE-4/survivin/ her2 /COX-2 CTL epitope peptides .

DETAILED DESCRIPTION:
All participants judged to have RCC and considered able to conduct apheresis. Immunotherapy regimen will include subcutaneous injection (3million cells) DC1 vaccines and intravenous infusion CTL cells. On day 0,participants conduct apheresis for 50-60ml. PBMCs were separated from paiticipants by density gradient centrifugation. The adherent cells were initiated into DC followed by the particular combination of cytokines to promote DC type-1 polarization. On day 6, the synthetic CTL epitope peptides were added into the culture for autologous DCs for another 24h. Then one half of DC1s were resuspended in 1ml normal saline for clinical multi-point injection near lymph nodes. The remaining half were cocultured with autologous T cells for another 7 days to induce antigen-specific CTL cells. The applied TAAs included MAGE-3/ MAGE-4/ survivin/ her2 /ect. On day 14, after quality inspection qualified, CTL cells were harvested and resuspended in 100ml normal saline and 2% autologous plasma for clinical intravenous infusion, once a day for 3 days. In order to avoid overlap between experimental immunotherapy and potential adjuvant chemotherapy, chemotherapy may start at least 2 weeks after completion of the cycle of immunotherapy. The 2nd cycle of immunotherapy may start at least 4weeks after the completion of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

Patients with histologically confirmed stage III-IV renal malignancies; The patient underwent radical operation of RCC within 8 weeks before enrollment; Must have normal marrow hematopoiesis function as defined below: Hemoglobin≥90g/L, WBC>4000/mm3, Absolute Neutrophil Count (ANC)≥1500/µL, Platelet≥ 100,000/µL, Must have normal important organ function as defined below: Total bilirubin≤1.5 x institutional upper limit of normal(ULN), AST(SGOT) and ALT(SGPT)≤2.5x ULN , ALP≤1.5x ULN; BUN and Creatinine <1.5x ULN, Creatinine clearance ≥80mL/min.

life expectancy≥3 months; No other serious heart, liver and kidney organ dysfunction; Quality of life score (Karnofsky performance score) ≥60; Patients must be able to understand and be willing to sign a written informed consent document.

Exclusion Criteria:

Prior allergic reaction or hypersensitivity to cytokines (eg.IL-2); Patients with systemic or local infection requiring anti-infectious treatment; Patients currently treated with systemic immunosuppressive agents, including steroids, Patients with active autoimmune disease or history of transplantation requiring steroid treatment; Tested positive for HIV; Pregnant or lactating women Patients with important organ dysfunction; Any reason that, in the opinion of the investigator, contraindicates that the patient participates in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 24 weeks
  Our primary objective is to evaluate whether our cellular therapy regimen is safe.

SECONDARY OUTCOMES:
G250 mRNA figures | 24 weeks

OTHER OUTCOMES:
T cell subsets figures | 12 weeks
Serum cytokine secretion figures | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Junnian Zheng, MD, Principal Investigator — Xuzhou Medical University

IPD SHARING:
Plan to Share IPD: No